CLINICAL TRIAL: NCT00811616
Title: Safety And Efficacy Evaluation of Sirolimus Eluting Supralimus-Core™ Stent at MAX DDHV Institute in the Treatment of de Novo Native Coronary Artery Lesions
Brief Title: A Safety and Efficacy of Supralimus™ Core™ Sirolimus Eluting Stent at MAX DDHV Institute
Acronym: Maximus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The MAXIMUS study
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Supralimus-Core™; de novo native coronary artery lesion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supralimus™ Core™ Sirolimus eluting stent (Experimental): Supralimus™ Core™ Sirolimus eluting stent manufactured by Sahajanand Medical Technologies Limited intended to treat coronary artery disease.
  Interventions: Device: Supralimus-Core™; Device: Supralimus™ Core™ Sirolimus eluting stent

INTERVENTIONS:
Device: Supralimus-Core™ — Sirolimus Eluting Cobalt Chromium based coronary stent system
Device: Supralimus™ Core™ Sirolimus eluting stent — Supralimus™ Core™ Sirolimus eluting stent intended to treat coronary artery disease.

SUMMARY:
OBJECTIVES:

The primary objective of this study is to assess the safety and efficacy of the Supralimus - Core™ Sirolimus Eluting Stent in de novo native vessel obstructive coronary artery disease.

STUDY DESIGN:

This is a single centre, prospective study. Approximately 105 patients were enrolled in the study. Patients were followed for twelve months post-procedure. All patients were to have a repeat angiography at 8 months.

STUDY POPULATION:

The study population consisted of approximately 105 patients with de novo native vessel obstructive coronary artery disease with no specific criteria. Patients from the daily practice were included. Patients had to meet all eligibility criteria for inclusion into the study.

ENDPOINTS:

The primary safety endpoint of the study is defined as Major Adverse Cardiac Events (MACE) at 30 days.

The primary efficacy endpoint is the in-stent binary restenosis rate at 8-month follow-up determined by off-line Quantitative Coronary Angiography.

The following secondary efficacy endpoints were assessed

* Angiographic success
* Procedure success
* Quantitative Coronary Angiography derived vessel parameters in-stent and 5 mm proximal and 5 mm distal from the edge of the stent: acute gain, MLD, % DS, late loss, mean diameter. In-stent pre-, post and at 8-month follow-up.
* Clinically justified Target Lesion Revascularization (TLR) at 12 months

The following secondary safety endpoints were assessed:

* MACE until 12 months
* Device related SAEs until 12 months
* Angiographic stent thrombosis: Subacute (after procedure until 30 days) and Late (after 30 days until 12 months)

ELIGIBILITY:
Inclusion Criteria:

* The patient must be >= 18 years of age;
* Symptomatic ischemic heart disease (CCS class 1 -4 , Braunwald class IB, IC, IIB, IIC, IIIB,IIIC) and/or objective evidence of myocardial ischemia;
* Vessel size of >= 2.5 and <= 3.5mm.
* Target lesions which can be covered by stent in a manner lesion stent ratio of at least 1.5.
* Acceptable candidate for coronary artery bypass surgery (CABG);
* Target lesion stenosis is >50% and <100% (TIMI flow I) (visual estimate);
* The patient has been informed of the nature of the study agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee (MEC) or Institutional Review Board (IRB).

Exclusion Criteria:

* Women of childbearing potential;
* Impaired renal function (creatinine > 2.0 mg/dl or 177 µmol/l);
* Any patient who has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis);
* Recipient of heart transplant;
* Restenotic or lesion in graft.
* Patient with a life expectancy less than 12 months;
* Known allergies to aspirin, clopidogrel bisulphate (Plavix), ticlopidine (Ticlid), heparin or stainless steel;
* Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in an investigational drug or another device study, or subject to inclusion in another investigational drug or another device study during follow-up.

Angiographic Exclusion criteria:

* Unprotected left main coronary artery disease with >=50% stenosis;
* Angiographic evidence of thrombus (thrombus larger than half the diameter of the vessel and/or requiring other interventions such as angiojet, exciser, thrombolysis, etc.);
* Ejection fraction <= 30%;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Primary safety endpoint: Major Adverse Cardiac Events (MACE) | 30 days
Primary efficacy endpoint: In-stent binary restenosis rate determined by off-line Quantitative Coronary Angiography. | 8 Month

SECONDARY OUTCOMES:
Secondary safety endpoints: - MACE until 12 months, Device related SAEs until 12 months, Angiographic stent thrombosis: Subacute (after procedure until 30 days) and Late (after 30 days until 12 months) | 12 months
Secondary efficacy endpoints: Angiographic, Procedure success; acute gain, MLD, % DS, LL, mean diameter; In-stent pre-,post,8-month follow-up; Clinically justified TLR at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ashok Seth, Principal Investigator — Escorts Heart Institute & Research Centre
Locations (1):
- Max Heart and Vascular Institute, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Seth A, Chandra P, Chouhan NS, Thakkar AS. A first-in-man study of sirolimus-eluting, biodegradable polymer coated cobalt chromium stent in real life patients. Indian Heart J. 2012 Nov-Dec;64(6):547-52. doi: 10.1016/j.ihj.2012.07.011. Epub 2012 Jul 27. PMID 23253405